CLINICAL TRIAL: NCT03608124
Title: Behavior Management Techniques Adopted by Pediatric Dentists in Egypt: Cross-sectional Study
Brief Title: Behavior Management Techniques Adopted by Pediatric Dentists in Egypt
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Samah Mohsen Kanzel, Samah Mohsen Omer Salem Kanzel, Cairo University
Other Study IDs: CEBD-CU-2018_06_18
Record Dates: First submitted 2018-07-14; First posted 2018-07-31 (Actual); Last update posted 2018-07-31 (Actual); Status verified 2018-07

CONDITIONS: Child Anxiety

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Behavior management techniques — Pediatric dentists will be questionnaired regarding their adopted behavior management techniques for pediatric patients

SUMMARY:
A cross-sectional study to investigate behavior management techniques used by pediatric dentists in Egypt according to AAPD clinical guidelines.

DETAILED DESCRIPTION:
Observational study to investigate behavior management techniques adopted by pediatric dentists in Egypts for different patients ages, by distributing questionnaires in Egyptian govermental universities consisting of participant's demographic information, behavior management techniques used for each age group and their opinion or comments.

ELIGIBILITY:
Inclusion Criteria:

* pediatric dentist and holding at least a master degree

Exclusion Criteria:

* refusal to participate

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Pediatric dentists either govermental university staff in Cairo or Phd students in Cairo govermental universities
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2017-07-01 (Actual); Study Completion 2017-08-15 (Actual)

PRIMARY OUTCOMES:
Behavior management | one month
  Questionnaire will be used for measurement using binary questions (Yes, No) to measure the outcome. Summing up Yes responses will reveal the most common behavior management techniques used by pediatric dentists in Egypt

CONTACTS AND LOCATIONS:
Overall Officials: Hassan A. Ahmed, ahmed, Study Director — Centre of evidence based dentistry
Locations (1):
- Cairo university, Giza, Manial, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
Protocol will be shared